CLINICAL TRIAL: NCT06509841
Title: The Impact of Jiaji Electroacupuncture and Scalp Electroacupuncture on Traumatic Spinal Cord Injury: A Randomized Controlled Trial
Brief Title: The Impact of Jiaji Electroacupuncture and Scalp Electroacupuncture on Traumatic Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202401
Record Dates: First submitted 2024-07-06; First posted 2024-07-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2022-07

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: spinal cord injury; electroacupuncture; Jiaji acupoint; scalp acupuncture; clinical efficacy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scalp electro-acupuncture (Experimental): Recruiting patients receiving electro-acupuncture at the Scalp points
  Interventions: Other: Electro-acupuncture at the scalp points
- Jiaji electro-acupuncture (Experimental): Recruited patients receiving electro-acupuncture at the Jiaji points
  Interventions: Other: Electro-acupuncture at the Jiaji points

INTERVENTIONS:
Other: Electro-acupuncture at the Jiaji points — Adopting treatments for the group that received electro-acupuncture at the Jiaji points, including: ① electro-acupuncture at the Jiaji points with continuous treatment for 8 weeks.
  Arms: Jiaji electro-acupuncture
Other: Electro-acupuncture at the scalp points — Adopting treatments for the group that received electro-acupuncture at the Scalp points, including: ① electro-acupuncture at the Scalp points with continuous treatment for 8 weeks.
  Arms: Scalp electro-acupuncture

SUMMARY:
Spinal cord injury (SCI), leads to functional deficits and complications like neurogenic bladder and deep vein thrombosis, imposing a global annual financial burden. This trial aims to compares Jiaji electroacupuncture (JEA) and scalp electroacupuncture (SEA) in SCI rehabilitation. This randomized controlled trial (RCT) compared JEA and SEA in SCI rehabilitation.

DETAILED DESCRIPTION:
The motor function score, light touch score, and pinprick sensation score of both groups showed significant improvement ( P < 0.001). When comparing Group A and Group B, there was no statistically significant difference in ASIA grade improvement at week 4 ( P > 0.05), but at week 8 and the 3-month follow-up, the proportion of ASIA grade improvement in Group A was significantly higher than that in Group B (week 8: 40.48% vs. 14.29%, P=0.007; 3-month follow-up: 47.62% vs. 21.43%, P = 0.012). At week 4, week 8, and the 3-month follow-up, Group A's motor function score, light touch score, pinprick sensation score, and MBI were all higher than those of Group B ( P < 0.05).

ELIGIBILITY:
Inclusion Criteria:

1. The duration of spinal cord injury must be between 3 to 6 months;
2. The site of injury must be clearly defined;
3. The cause of injury must be traumatic;
4. Patients must be over 18 years of age;
5. Patients must provide consent to participate in this study.

Exclusion Criteria:

1. Unknown time or site of injury;
2. Disagreement to participate in this study;
3. Patients with contraindications for acupuncture intervention (such as skin lesions or rashes at potential acupuncture sites);
4. Patients with cognitive or language impairments who are unable to cooperate with scale evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
ASIA Score | 0 week, 4 weeks, 8 weeks, and 3 months of follow-up (3 months after the end of treatment)
  The ASIA score for spinal cord injury, established by the American Spinal Injury Association, serves as a method to assess the severity of spinal cord injuries and functional recovery. It includes evaluations of the patient's neurological motor function, light touch sensation score, pinprick sensation score, and sphincter function performance. The ASIA score categorizes spinal cord injuries into five grades: 1/A, 2/B, 3/C, 4/D, and 5/E. A lower grade indicates a more severe injury, characterized by weaker motor and sensory scores, including light touch and pinprick sensation scores.
Modified Barthel Index | 0 week, 4 weeks, 8 weeks, and 3 months of follow-up (3 months after the end of treatment)
  The Modified Barthel Index Rating Scale is a tool used to assess adults' abilities to perform activities of daily living. It comprises 10 assessment items, including feeding, bathing, grooming, dressing, and controlling bowel and bladder movements. Each item is divided into different levels corresponding to various scores, with a maximum score of 100. A score of ≥60 indicates mild functional impairment, a score of 59-41 indicates moderate functional impairment, and a score of ≤40 indicates severe functional impairment.
Incidence of Complications | 0 week, 4 weeks, 8 weeks, and 3 months of follow-up (3 months after the end of treatment)
  Monitor whether patients experience severe bleeding, pressure ulcers, deep vein thrombosis, neurogenic bowel dysfunction, neurogenic bladder, nephropathy, pulmonary infections, traumatic encephalopathy, pain, and other complications during the treatment and follow-up periods. Record the number of patients with each type of complication. The incidence rate of complications is calculated as follows: (Total number of cases with a specific complication in each group) ÷ (Total number of patients in that group) × 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Zhejiang Provincial People's Hospital to Hangzhou Medical College., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucci VM, McGrath MS, Inskip JA, Sarveswaran S, Willms R, Claydon VE. Clinical recommendations for use of lidocaine lubricant during bowel care after spinal cord injury prolong care routines and worsen autonomic dysreflexia: results from a randomised clinical trial. Spinal Cord. 2020 Apr;58(4):430-440. doi: 10.1038/s41393-019-0381-2. Epub 2019 Nov 25. PMID 31767947
- [Background] Dyson-Hudson TA, Kadar P, LaFountaine M, Emmons R, Kirshblum SC, Tulsky D, Komaroff E. Acupuncture for chronic shoulder pain in persons with spinal cord injury: a small-scale clinical trial. Arch Phys Med Rehabil. 2007 Oct;88(10):1276-83. doi: 10.1016/j.apmr.2007.06.014. PMID 17908569
- [Background] Xiong F, Fu C, Zhang Q, Peng L, Liang Z, Chen L, He C, Wei Q. The Effect of Different Acupuncture Therapies on Neurological Recovery in Spinal Cord Injury: A Systematic Review and Network Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2019 Oct 27;2019:2371084. doi: 10.1155/2019/2371084. eCollection 2019. PMID 31772592
- [Background] Tang H, Guo Y, Zhao Y, Wang S, Wang J, Li W, Qin S, Gong Y, Fan W, Chen Z, Guo Y, Xu Z, Fang Y. Effects and Mechanisms of Acupuncture Combined with Mesenchymal Stem Cell Transplantation on Neural Recovery after Spinal Cord Injury: Progress and Prospects. Neural Plast. 2020 Sep 25;2020:8890655. doi: 10.1155/2020/8890655. eCollection 2020. PMID 33061954
- [Background] Xiong F, Lu J, Pan H, Wang F, Huang Y, Liu Y, Li L, Zhang R, Wang Y, He C, Quan W. Effect of Specific Acupuncture Therapy Combined with Rehabilitation Training on Incomplete Spinal Cord Injury: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2021 Dec 26;2021:5671998. doi: 10.1155/2021/5671998. eCollection 2021. PMID 34987595
- [Background] Jiang K, Sun Y, Chen X. Mechanism Underlying Acupuncture Therapy in Spinal Cord Injury: A Narrative Overview of Preclinical Studies. Front Pharmacol. 2022 Apr 7;13:875103. doi: 10.3389/fphar.2022.875103. eCollection 2022. PMID 35462893
- [Background] Huang Y, He K, Fang D, Ni F, Qiu B, Liang K, Ma R. A bibliometric of research trends in acupuncture for spinal cord injury: Quantitative and qualitative analyses. Front Neurol. 2022 Sep 15;13:936744. doi: 10.3389/fneur.2022.936744. eCollection 2022. PMID 36188361
- [Background] Fan Q, Cavus O, Xiong L, Xia Y. Spinal Cord Injury: How Could Acupuncture Help? J Acupunct Meridian Stud. 2018 Aug;11(4):124-132. doi: 10.1016/j.jams.2018.05.002. Epub 2018 May 30. PMID 29753705
- [Background] Inzani F, Rindi G. Introduction to neuroendocrine neoplasms of the digestive system: definition and classification. Pathologica. 2021 Feb;113(1):1-4. doi: 10.32074/1591-951X-227. PMID 33686304